CLINICAL TRIAL: NCT04447664
Title: Telespirometry: Home Monitoring of Asthmatic Patients With Spirometer
Brief Title: Telemonitoring of Lung Function by Spirometry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TMED_SPIRO_001
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-03

CONDITIONS: Asthma in Children; Asthma
Keywords: Spirometry
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine arm (Experimental)
  Interventions: Device: Inclouded telespirometry system
- Control arm (No Intervention)

INTERVENTIONS:
Device: Inclouded telespirometry system — Components of the system: Portable digital ultrasonic spirometer (Uscom SpiroSonic MOBILE), android mobile application, clinical web cloud application
  Arms: Telemedicine arm

SUMMARY:
Asthma is the most common respiratory disorder in children that causes breathing problems. The patients may have respiratory symptoms such as cough, wheeze, or short of breath. Asthma can be mild or severe when daily activities become compromised. Generally, by application of proper treatment, asthma symptoms can be well controlled. However, the exacerbation of the disease often leads to acute respiratory adverse events that require hospitalization and school absenteeism.

In this study, we plan the remote monitoring of lung function parameters in asthmatic children (under 18 years of age). We hypothesize that the daily home monitoring of respiratory indices will predict the occurrence of exacerbation and the hospitalization can be lowered.

Asthmatic children arriving for the regular examinations to the Department of Pediatrics and Pediatric Health Care Center of the University of Szeged will be involved. The patients are randomly divided into two treatment groups, telemonitoring and control.

For both groups, general patient characteristics will be recorded, and lung function parameters will be measured with a clinical spirometer.

Patients in the telemedicine group receive the home mobile controlled spirometer and trained by a pediatric pulmonologist for home examination. The spirometers are handed for 12 months, and children are asked to perform measurements minimum 4 times per week (at least one day a week in the morning and in the evening). In the case of asthma attacks, more frequent measurements repeated several times a day are required. Children in the telemedicine group complete the Asthma Control Test (ACT) after each measurement, which provides a numerical score related to the severity of asthma symptoms. Lung function parameters measured by children and the ACT results are automatically uploaded to a clinical server where the pulmonologists and built-in algorithms are monitoring the quality of the data. In case of deterioration of the lung function parameters, the patients are called for a personal visit and their treatment can be revised.

Every three months, members of both groups come to the outpatient clinic for a personal visit, where the same examinations are performed.

DETAILED DESCRIPTION:
Asthma is the most common respiratory disorder in children characterized by periodic airway obstruction, bronchial hyper-responsiveness, and airway inflammation. The symptoms of asthma may include cough, wheeze, or bronchoconstriction with airflow limitation. The severity of asthma may vary from mild to severe. Mild asthma is associated with rear events of short of breath. However, the exacerbation of the disease often leads to acute respiratory adverse events with severe hypoxia that requires hospitalization. The hospital care involves travel costs for the children and parents, school and work absenteeism.

The primary objective of the study is to investigate whether the annual occurrence of asthma exacerbation can be decreased by the use of the telespirometry system. Another objective is to determine which lung function parameters are best to predict asthma exacerbation.

To address these aims we plan to involve two groups (telemonitoring and control) of asthmatic children with GINA 2-5 stage under 18 years of age. Poor general condition, any disease which endangers the health of the volunteer or contraindicates the study and lack of parental consent are defined as the exclusion criteria.

The lung function in the children in both groups will be monitored by conventional spirometric assessment performed at the Department of Pediatrics and Pediatric Health Care Center of the University of Szeged. After each lung function assessments children will be asked to fill the Asthma Control Test (ACT).

Patients in the telemedicine group receive the home mobile controlled spirometer and trained by a pediatric pulmonologist for home examination. The spirometers are handed for 12 months, and children are asked to perform measurements minimum 4 times per week (at least one day a week in the morning and in the evening). In the case of asthma exacerbation, more frequent measurements repeated several times a day are required. Children in the telemedicine group complete the ACT after each measurement, which provides a numerical score related to the severity of asthma symptoms. Lung function parameters measured by children and the ACT test results are automatically uploaded to a clinical server where the pulmonologists and built-in algorithms are monitoring the quality of the data. In case of deterioration of the lung function parameters, the patients are called for a personal visit and their treatment can be revised.

Every three months, members of both groups come to the outpatient clinic for a personal visit, where the same examinations are performed.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 18 years
* signed ICF
* asthmatic children with 2-5 GINA score
* The children is open-minded for telespirometric measurements at home and is capable for those measurements
* Parent understands and supports the investigation

Exclusion Criteria:

* Withdrawal of consent
* Any disease which, by the investigators opinion, is a risk for the patients health and/or is contraindicating the participation in the study
* Bad general condition

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of asthma exacerbations per year | 12 months
  Change of the incidence of asthma exacerbations per year using telespirometry system

SECONDARY OUTCOMES:
expiratory Forced Vital Capacity (FVC), the maximum amount of air that can forcibly be blown out after full inspiration | 12 months
  Lung function parameters to predict asthma exacerbation
Forced Expiratory Volume in one second (FEV1), is the volume of air that can forcibly be blown out in first 1 second after full inspiration | 12 months
  Lung function parameters to predict asthma exacerbation
FEV1/FVC ratio (FEV1%) | 12 months
  Lung function parameters to predict asthma exacerbation
Peak Expiratory Flow (PEF), peak expiratory flow rate during expiration | 12 months
  Lung function parameters to predict asthma exacerbation
Forced Expiratory Flow at 25-75% of FVC (FEF25-75%), mean of forced expiratory flow over the middle half of the FVC | 12 months
  Lung function parameters to predict asthma exacerbation
The change of absenteeism days from work/school | 12 months
  Effect of the use of telemedicinal system for the asthma control

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No